CLINICAL TRIAL: NCT02616042
Title: The Effect of New Dentifrices Containing Centella Asiatica and Bamboo Salt on Reducing Plaque and Gingivitis: a Randomized Clinical Trial
Brief Title: The Effect of New Dentifrices Containing Centella Asiatica and Bamboo Salt on Reducing Plaque and Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Household & Health Care Ltd. (Industry)
Collaborators: Seoul National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRI09001
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Labor Trial Refused
Keywords: Centella asiatica; bamboo salt; dentifrice
MeSH Terms: interventions — Centella asiatica extract; bamboo salt

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Centella asiatica and bamboo salt (Experimental): Participants received a dentifrice which contains Centella asiatica, bamboo salt, dental-type silica, sodium fluoride and aminocaproic acid. Each participant brushed their teeth using only the assigned dentifrices for 3 minutes twice a day (after breakfast and before bedtime). All participants used the assigned dentifrices for 4 days in each trial cycle.
  Interventions: Other: Centella asiatica and bamboo salt; Other: Centella asiatica
- Centella asiatica (Experimental): Participants received a dentifrice which contains Centella asiatica, dental-type silica, sodium fluoride and aminocaproic acid. Each participant brushed their teeth using only the assigned dentifrices for 3 minutes twice a day (after breakfast and before bedtime).
  Interventions: Other: Centella asiatica and bamboo salt; Other: Centella asiatica
- Control dentifrice (Placebo Comparator): Participants received a plain dentifrice which contains dental-type silica, sodium fluoride and aminocaproic acid. Each participant brushed their teeth using only the assigned dentifrices for 3 minutes twice a day (after breakfast and before bedtime).
  Interventions: Other: Centella asiatica and bamboo salt; Other: Centella asiatica

INTERVENTIONS:
Other: Centella asiatica and bamboo salt — Participants uses three types of dentifrices for four days after each wash-out period of 10 days. Dentifrice with Centella asiatica and bamboo salt is compared with control dentifrice.
Other: Centella asiatica — Participants uses three types of dentifrices for four days after each wash-out period of 10 days. Dentifrice with Centella asiatica is compared with control dentifrice.

SUMMARY:
This study aims to evaluate the effect of dentifrice formulations containing Centella asiatica and bamboo salt on gingivitis and dental plaque. Participants uses dentifrice which contains Centella asiatica and bamboo salt and the same participants will also use placebo for tooth brushing by cross-over design.

DETAILED DESCRIPTION:
With growing interest in plant-based products among researchers, many toothpastes with various herbal extracts have been introduced over the past few decades,Centella asiatica (CA), a small herb broadly cultivated in China, Southeast Asia, India and Oceanic countries, has long been used for therapeutic purposes since ancient times.CA has been reported to be useful in the treatment of skin diseases wound repair and healing of burn. In dentistry, few studies have explored the efficacy of CA. In one study, CA was demonstrated to be an effective supportive agent following periodontal treatment, resulting in reduced plaque and gingivitis. In spite of such wound healing properties of CA, its usage in dental field has been limited.

Bamboo salt (BS) is a Korean folk remedy consisting of sea salt roasted in bamboo which has long been used for therapeutic purposes in Korea. Toothpastes containing BS has been sold in Korea for some decades. Some in vitro studies and animal studies using rats demonstrated anti-inflammatory effects of BS. Nevertheless, no human study has yet evaluated the effect of BS on periodontal health.

Therefore, the new dentifrice containing CA and BS was developed.

ELIGIBILITY:
Inclusion Criteria:

* Systemical healthy individual
* Normal alignment of teeth

Exclusion Criteria:

* Recent antibiotic treatment
* Existence of dental caries or periodontitis
* Those needs emergency dental treatments
* Natural teeth less than 20
* Denture wearer
* Oral appliance for orthodontic treatment
* Pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Gingivitis | Four day
  Gingival index is measured

SECONDARY OUTCOMES:
Dental plaque | Four day
  Plaque index is measured

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Duck Kim, DDS, PhD, Principal Investigator — Seoul National University